CLINICAL TRIAL: NCT05810766
Title: Effects of Mobilization With Movement Techniques of Shoulder Girdle on Pain, Range of Motion and Function in Patients With Chronic Adhesive Capsulitis
Brief Title: Mobilization With Movement Techniques of Shoulder Girdle in Patients With Chronic Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0115
Record Dates: First submitted 2023-03-08; First posted 2023-04-12 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive Capsulitis; Manual therapy; Mobilization therapy
MeSH Terms: conditions — Bursitis | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization with movement Group (Experimental): Week 1 & 2: mobilization with movement at glenohumeral joint for improving flexion, abduction internal and external rotation. 3 sets of painless glides of 10 repetitions will be given, with 1 minute rest between sets.
  * Week 2 & 4:MWM at glenohumeral joint and then we will add progression by adding glides at sternoclavicular and acromioclavicular joint.5 sets of painless glides of 10 repetitions will be given, with 3-minute rest between sets.
  * Week 3 & 6:MWM at glenohumeral joint and glides at sternoclavicular, acromioclavicular along with glides at scapulothoracic. 5 sets of painless glides for 10 repetitions were given. Progression can be introduced by increasing the number of repetitions performed exercises for 3 weeks.
  Interventions: Other: mobilization with movement
- conventional physical therapy (Other): Hot pack for 15 minutes
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: mobilization with movement — MWM at glenohumeral joint and then we will add progression by adding glides at sternoclavicular and acromioclavicular joint.5 sets of painless glides of 10 repetitions will be given, with 3-minute rest between sets.
  Arms: mobilization with movement Group
Other: conventional physical therapy — Hot pack for 15 minutes
  Arms: conventional physical therapy

SUMMARY:
Study will be a Randomized clinical trial to check Effects of mobilization with movement techniques of shoulder girdle on pain, range of motion and function in patients with chronic adhesive capsulitis so that we can devise a treatment protocol Total Thirty subjects will be included in this study .Out of total 15 will be randomly allocated via lottery method in group 1 and 15 will be allocated in group 2. Group 1 will receive hot packs for 15 minutes for warming up, shoulder girdle mobilization with movement techniques along with other shoulder girdle joints mobilizations (sternoclavicular, acromioclavicular, cervicothoracic and scapulothoracic joints) and conventional physical therapy treatment while group 2 will receive only hot pack for 15 minutes and conventional physical therapy management. All patients will be treated for 12 sessions, two sessions per week for 6 weeks. Shoulder pain and disability index consist of two parts, part one which assesses pain severity and part two which assesses functional disability. Study setting will be suraiya majeed trust hospital. Assessment will be done at 0 weeks, 3 weeks, and 6 weeks. Data was analysed by using SPSS version 26.

DETAILED DESCRIPTION:
The term "adhesive capsulitis describes the condition in which there is a restriction of active and passive ranges of the shoulder joint due to the thickening of the synovial capsule, pain, and stiffness. Our ability to interact with our surroundings is made possible by the shoulder's exceptional range of motion (ROM), which makes it a special anatomical structure. This study aims to determine the effects of mobilization with movement techniques of shoulder girdle on pain, range of motion, and function in patients with chronic adhesive capsulitis. Patients of both genders, idiopathic adhesive capsulitis, age group between 25-55 years, minimum six weeks chronicity of adhesive capsulitis, and patients with positive Apley's scratch test for adhesive capsulitis will be included, Patients having bilateral adhesive capsulitis, fractures of the Shoulder girdle, Rheumatoid arthritis/ osteoarthritis, severe joint pain unrelieved by rest and any bony or soft tissue systemic disease will be excluded In the previous literature there is study gap that provides a comprehensive treatment strategy for patients having chronic adhesive capsulitis The aim of this study is to apply MWM in patients having chronic adhesive capsulitis. A regional interdependence approach to shoulder dysfunction will be used in the treatment plan, taking into account the fact that glenohumeral function depends on scapular function, which in turn can also be affected by upper kinetic chain segments depending upon the patient's presentation, because of the close relation of surrounding joints (sternoclavicular, acromioclavicular, and scapulothoracic joints) with glenohumeral joint to gain complete effective shoulder ranges. That is why there is a great need for this study and in previous studies primarily acute patients were included therefore now it is necessary to draw attention to chronicity in adhesive capsulitis patients.

Mobilization with movement at the glenohumeral joint for improving flexion, abduction internal and external rotation. 3 sets of painless glides of 10 repetitions were given, with 1-minute rest between sets. and progression was added

Both groups received hot packs for 15 minutes for warming up and conventional physical therapy treatment

ELIGIBILITY:
Inclusion Criteria:

* • Patients of Both gender

  * Age 25-55 years
  * Minimum 6 weeks chronicity of adhesive capsulitis
  * Positive Apley's scratch test for adhesive capsulitis
  * Idiopathic adhesive capsulitis

Exclusion Criteria:

* • Bilateral adhesive capsulitis

  * Fractures of the Shoulder girdle
  * Rheumatoid arthritis/ osteoarthritis
  * Severe joint pain unrelieved by rest.
  * Any bony or soft tissue systemic disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | up to 6 weeks
  Patients are asked to circle the number on a Numerical Rating Scale (NRS) that best describes their level of discomfort between 0 and 10, 0 and 20, or 0 and 100. The lower limit often denotes "the least amount of suffering ," whereas zero typically denotes "no pain at all."
Goniometer | up to 6 weeks
  The most popular and reliable approach for determining shoulder range of motion (ROM) is by utilizing a goniometer. A goniometer is a straightforward instrument that has two arms joined at a hinge. The goniometer's second arm would be used to measure the joint angle while the physiotherapist placed one arm of the patient against the patient's body
Shoulder pain and disability index (SPADI) | up to 6 weeks
  The Shoulder Discomfort and Disability Index is a tool that may be used to determine the level of pain in people with adhesive capsulitis (SPADI). It was created to assess current shoulder discomfort and impairment in outpatients.(9) The Shoulder Pain and Disability Index (SPADI), a patient-completed questionnaire of 13 items, measures the severity of pain and the degree to which daily activities involving the use of the upper extremities are made more difficult. There are 5 items on the pain subscale and 8 on the disability subscale.

CONTACTS AND LOCATIONS:
Overall Officials: khadija Musarat, MS*, Principal Investigator — Riphah International University
Locations (1):
- Suraiya majeed trust hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manske RC, Prohaska D. Diagnosis and management of adhesive capsulitis. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):180-9. doi: 10.1007/s12178-008-9031-6. PMID 19468904
- [Background] Ramirez J. Adhesive Capsulitis: Diagnosis and Management. Am Fam Physician. 2019 Mar 1;99(5):297-300. PMID 30811157
- [Background] Nakandala P, Nanayakkara I, Wadugodapitiya S, Gawarammana I. The efficacy of physiotherapy interventions in the treatment of adhesive capsulitis: A systematic review. J Back Musculoskelet Rehabil. 2021;34(2):195-205. doi: 10.3233/BMR-200186. PMID 33185587
- [Background] Patel R, Urits I, Wolf J, Murthy A, Cornett EM, Jones MR, Ngo AL, Manchikanti L, Kaye AD, Viswanath O. A Comprehensive Update of Adhesive Capsulitis and Minimally Invasive Treatment Options. Psychopharmacol Bull. 2020 Oct 15;50(4 Suppl 1):91-107. doi: 10.64719/pb.4384. PMID 33633420
- [Background] Georgiannos D, Markopoulos G, Devetzi E, Bisbinas I. Adhesive Capsulitis of the Shoulder. Is there Consensus Regarding the Treatment? A Comprehensive Review. Open Orthop J. 2017 Feb 28;11:65-76. doi: 10.2174/1874325001711010065. eCollection 2017. PMID 28400876
- [Background] Doner G, Guven Z, Atalay A, Celiker R. Evalution of Mulligan's technique for adhesive capsulitis of the shoulder. J Rehabil Med. 2013 Jan;45(1):87-91. doi: 10.2340/16501977-1064. PMID 23037929
- [Background] Ali SA, Khan M. Comparison for efficacy of general exercises with and without mobilization therapy for the management of adhesive capsulitis of shoulder - An interventional study. Pak J Med Sci. 2015 Nov-Dec;31(6):1372-6. doi: 10.12669/pjms.316.7909. PMID 26870099